CLINICAL TRIAL: NCT01979276
Title: A Phase I/II Study of Pomalidomide (CC-4047®), Dexamethasone and Romidepsin in Patients With Relapsed or Refractory Multiple Myeloma (Romi Poma)
Brief Title: Study of Pomalidomide, Dexamethasone, and Romidepsin for Rel/Ref Myeloma
Acronym: Romi Poma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: this study was terminated due to losing financial support, and enrollment challenges
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1306014005
Record Dates: First submitted 2013-10-25; First posted 2013-11-08 (Estimated); Results first posted 2018-01-31 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-05

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — romidepsin; pomalidomide; Dexamethasone

ARMS (1):
- Pomalidomide, Romidepsin, Dexamethasone (Experimental): Pomalidomide, 4 mg by mouth daily on days 1-21 of 28 day cycle Dexamethasone, 40 mg by mouth on days 1, 8, 15, and 22 of 28 day cycle Romidepsin, IV on days 1 and 15 of 28 day cycle, dose level to be determined Dexamethasone
  Interventions: Drug: Romidepsin; Drug: pomalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Romidepsin — Romidepsin intravenously on days 1 and 15 of a 28-day cycle
Drug: pomalidomide — Pomalidomide 4mg daily by mouth on days 1-21 of a 28-day cycle
Drug: Dexamethasone — Dexamethasone 40mg by mouth on days 1, 8, 15 and 22 of a 28-day cycle

SUMMARY:
This clinical trial is for subjects with multiple myeloma that has returned after treatment (relapsed) or did not respond to prior treatment (refractory). The study is in two parts, Phase I and Phase II. Phase I will determine the maximum tolerated dose of romidepsin in combination with pomalidomide and dexamethasone. The purpose of Phase II is to evaluate the effectiveness of combining romidepsin with pomalidomide and dexamethasone. The hypothesis is that overall response in a cohort of patients treated with romidepsin + pomalidomide + dexamethasone will be 60 percent.

DETAILED DESCRIPTION:
This phase I/II study is a treatment program for patients with relapsed or refractory multiple myeloma. Up to 48 patients will be enrolled. Phase I will follow a 3+3 dose escalation design to find the maximum tolerated dose of romidepsin in combination with pomalidomide and dexamethasone.

In Phase I, subjects will receive:

* Pomalidomide 4mg daily by mouth on days 1-21 of a 28-day cycle
* Dexamethasone 40mg by mouth on days 1, 8, 15 and 22 of a 28-day cycle
* Romidepsin intravenously (9 mg/m2, 12 mg/m2, 15 mg/m2 or 18 mg/m2) on days 1 and 15 of a 28-day cycle.

Phase II will expand the number of subjects in the MTD arm of the trial until 48 subjects are enrolled. In Phase II, subjects subjects will receive:

* Pomalidomide 4mg daily by mouth on days 1-21 of a 28-day cycle
* Dexamethasone 40mg by mouth on days 1, 8, 15 and 22 of a 28-day cycle
* Romidepsin intravenously on days 1 and 15 of a 28-day cycle at the Maximum Tolerated Dose determined by Phase I

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed multiple myeloma.
* measurable disease as defined by > 0.5 g/dL serum monoclonal protein, >0.1 g/dL serum free light chains, >0.2 g/24 hrs urinary M-protein excretion, and/or measurable plasmacytoma(s).
* relapsed or refractory multiple myeloma as defined by progression of disease either after prior therapy or lack of response to currently used therapy
* relapsed or progressive disease after at least 3 prior therapeutic treatments or regimens for multiple myeloma.
* refractory to bortezomib and lenalidomide
* >18 years at the time of signing the informed consent form.
* life expectancy of > 3 months.
* Karnofsky performance status > 70%, or > 60% if due to bony involvement of multiple myeloma
* normal organ and marrow function as defined below:

  1. Absolute Neutrophil Count > 1,000 cells/mm3 for Phase I, > 750 cells/mm3 for Phase II
  2. Platelet Count > 75,000/mm3 for Phase I, > 50, 000/mm3 for Phase II
  3. AST/ Serum SGOT < 3.0 x upper limits of normal
  4. ALT/ Serum SGPT < 3.0 x upper limit of normal
  5. Serum creatinine < 2.0 mg/dL
  6. Serum total bilirubin < 1.5 x upper limit of normal
* Laboratory test results within these ranges:

  g. Serum potassium ≥ 3.8 mmol/L h. Serum magnesium >1.8 mg/dL
* Females of child bearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL within 10-14 days prior to start of study drug(s) and again with 24 hours of prescribing pomalidomide (prescriptions must be filled within 7 days).
* Females of child bearing potential must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 4 weeks before starting pomalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with females of child bearing potential even if they have had a successful vasectomy.
* able to take aspirin (81 or 325 mg) daily as prophylactic anticoagulation (patients intolerant to ASA may use warfarin or low molecular weight heparin).
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Subjects with non-secretory Multiple Myeloma (no measurable monoclonal protein or plasmacytoma(s), free light chains, and/or M-spike in blood or urine).
* Patients with a prior history of other malignancies (except for basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix or breast) unless disease free for ≥ 3 years.
* Any known cardiac abnormalities such as:

  1. Congenital long QT syndrome
  2. QTc interval ≥ 480 milliseconds
  3. Myocardial infarction within 6 months of C1D1. Subjects with a history of myocardial infarction between 6 and 12 months prior to C1D1 who are asymptomatic and have had a negative cardiac risk assessment (treadmill stress test, nuclear medicine stress test, or stress echocardiogram) since the event may participate
  4. Other significant ECG abnormalities including 2nd degree atrio-ventricular (AV) block type II, 3rd degree AV block, or bradycardia (ventricular rate less than 50 beats/min)
  5. Symptomatic coronary artery disease (CAD), e.g., angina Canadian Class II-IV. In any subject in whom there is doubt, the subject should have a stress imaging study and, if abnormal, angiography to define whether or not CAD is present
  6. An ECG recorded at screening showing evidence of cardiac ischemia (ST depression depression of ≥2 mm, measured from isoelectric line to the ST segment). If in any doubt, the patient should have a stress imaging study and, if abnormal, angiography to define whether or not CAD is present
  7. Congestive heart failure (CHF) that meets New York Heart Association (NYHA) Class II to IV definitions (see Appendix E) and/or ejection fraction <40% by MUGA scan or <50% by echocardiogram and/or MRI;
  8. A known history of sustained ventricular tachycardia (VT), ventricular fibrillation (VF), Torsade de Pointes, or cardiac arrest unless currently addressed with an automatic implantable cardioverter defibrillator (AICD);
  9. Hypertrophic cardiomegaly or restrictive cardiomyopathy from prior treatment or other causes;
  10. Uncontrolled hypertension, i.e., blood pressure (BP) of ≥160/95; patients who have a history of hypertension controlled by medication must be on a stable dose (for at least one month) and meet all other inclusion criteria; or
  11. Any cardiac arrhythmia requiring an anti-arrhythmic medication (excluding stable doses of beta-blockers)
* Any Known seropositivity for or active viral infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV). Patients who are seropositive because of hepatitis B virus vaccine are eligible.
* Any active viral or bacterial infections or any coexisting medical problem that would significantly increase the risks of this treatment program.
* Any coexisting medical problem or laboratory evaluation that, in the treating physician's or principal investigator's opinion, makes the patient unsuitable to participate in this clinical trial.
* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
* Pregnant or breast feeding females. (Lactating females must agree not to breast feed while taking pomalidomide.)
* Subjects with any condition, including the presence of laboratory abnormalities, which in the opinion of the Investigator places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
* Use of any other experimental drug or therapy within 14 days of baseline.
* Subjects with a history of development of erythema nodosum, if characterized by a desquamating rash, while taking thalidomide, lenalidomide, pomalidomide or similar drugs.
* Concurrent use of other anti-cancer agents or treatment.
* Concomitant use of CYP3A4 inhibitors (See Appendix D)
* Prior therapy with romidepsin, thalidomide or pomalidomide
* Central nervous system or meningeal involvement
* Patients taking drugs leading to significant QT prolongation
* Known hypersensitivity to thalidomide or lenalidomide

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ruben Niesvizky, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two subjects were ineligible and therefore never started treatment.
Groups:
- ALL Patients: Pomalidomide, 4 mg by mouth daily on days 1-21 of 28 day cycle Dexamethasone, 40 mg by mouth on days 1, 8, 15, and 22 of 28 day cycle Romidepsin, IV on days 1 and 15 of 28 day cycle, dose level to be determined (9mg/m2, 12 mg/m2, 15 mg/m2 or 18 mg/m2)
Period: Overall Study
Arm/Group | ALL Patients
Started | 2
Completed (Completion defined as those removed from treatment due to disease progression (per protocol)) | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- ALL Patients: Pomalidomide, 4 mg by mouth daily on days 1-21 of 28 day cycle Dexamethasone, 40 mg by mouth on days 1, 8, 15, and 22 of 28 day cycle Romidepsin, IV on days 1 and 15 of 28 day cycle, dose level to be determined
Arm/Group | ALL Patients
Number analyzed (Participants) | 2
Age, Continuous [Mean (Full Range); unit: years] | 60.5 [58 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Number of Prior lines of therapy [Mean (Full Range); unit: Line of Prior Therapy] | 2.5 [2 to 3]
Beta 2 Microglobulin [Mean (Full Range); unit: mg/L] | 2.15 [2 to 2.3]
Lactate Dehydrogenase [Mean (Full Range); unit: U/L] | 209.5 [181 to 238]

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Romidepsin in Combination With Pomalidomide and Dexamethasone
Description: Establish a maximum tolerated dose (MTD) of romidepsin in combination with pomalidomide and dexamethasone in patients with relapsed or refractory multiple myeloma (phase I)
Time Frame: During the duration of the study (from first to last dose of study drug, on average ten 28-day cycles)
Population: MTD not established as study terminated while only 2 subjects enrolled. Only romidepsin dose tested was 9mg/mg2
Arm/Group | ALL Patients
Number analyzed (Participants) | 0

2. Primary Outcome: Efficacy of Study Regimen Combination
Description: The efficacy (as assessed by clinical response) of the combination of pomalidomide (CC-4047®) and romidepsin as therapy for patients with relapsed or refractory multiple myeloma (MM) (phase II portion) was evaluated using the IMWG Response Criteria for disease assessment. The best response was reported. (Criteria can be found at the following link, due to length and complexity of the response criteria: http://imwg.myeloma.org/international-myeloma-working-group-imwg-uniform-response-criteria-for-multiple-myeloma/)
Time Frame: From baseline to cycle of maximum response, which occurred on average after 2 cycles; 1 cycle = 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | ALL Patients
Number analyzed (Participants) | 2
Participants
  Progression of Disease | 1
  Very Good Partial Response | 1

3. Secondary Outcome: Time to Disease Progression (Progression Free Survival)
Time Frame: From start of treatment, to date of disease progression (on average, ten 28-day cycles)
Measure: Mean (Full Range); unit: cycles (defined as 28 days)
Arm/Group | ALL Patients
Number analyzed (Participants) | 2
cycles (defined as 28 days) | 9.5 [1 to 18]

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from baseline until removal from study. Serious adverse events were recorded from baseline until 30 days after the last dose of study drug.
Description: Adverse events were recorded using the CTCAE version 4.0. Serious adverse events were recorded from baseline until 30 days after the last dose of study drug.
Arm/Group | Pomalidomide, Romidepsin, Dexamethasone
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pomalidomide, Romidepsin, Dexamethasone (N=2)
Insomnia (Psychiatric disorders) | 1 (4)
Dyspnea with moderate exertion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Peripheral Neuropathy (Nervous system disorders) | 1 (1)
Blurred Vision (Eye disorders) | 1 (2)
Nausea - intermittent (Gastrointestinal disorders) | 1 (2)
Nausea (Gastrointestinal disorders) | 1 (3)
Dyspepsia - intermittent (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Generalized weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
constipation (Gastrointestinal disorders) | 1 (1)
Paresthesia around mouth (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (4)
Palpitations (Cardiac disorders) | 1 (2)
upper respiratory infection (Infections and infestations) | 1 (2)
tremors (Nervous system disorders) | 1 (2)
agitation (Psychiatric disorders) | 1 (1)
bloating (Gastrointestinal disorders) | 1 (1)
Stomach pain - epigastric area (Gastrointestinal disorders) | 1 (1)
ear infection (Infections and infestations) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2)
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (4)
urinary tract infection (Infections and infestations) | 1 (2)
pain - bilateral hips (General disorders) | 1 (2)
ALT elevation (Hepatobiliary disorders) | 1 (5)
AST elevation (Hepatobiliary disorders) | 1 (2)
headache (Nervous system disorders) | 1 (1)
nail infection (Infections and infestations) | 1 (1)
jaw pain (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less